CLINICAL TRIAL: NCT04427592
Title: Placenta Accreta; A Vision for Conservative Surgery
Brief Title: New Conservative Technique for Placenta Accreta Spectrum
Acronym: percreta
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Alexandria University (Other)
Responsible Party: Principal Investigator, Mahmoud A Hamdy, principal investigator, Alexandria University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: H.R501
Record Dates: First submitted 2020-05-31; First posted 2020-06-11 (Actual); Last update posted 2023-12-06 (Actual); Status verified 2023-12

CONDITIONS: Placenta Accreta Spectrum
MeSH Terms: conditions — Placenta Accreta | interventions — Ultrasonography

STUDY DESIGN:
Intervention Model Description: Investigators conducting prospective study for management of placenta accreta spectrum including diagnosis and uterine sparing surgery.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- pregnant women with placenta accreta spectrum (Experimental): The participants were subjected to ultrasound to diagnose placenta accreta spectrum followed by new conservative surgical technique.
  Interventions: Diagnostic Test: ultrasound; Procedure: closure of uterine wall defect

INTERVENTIONS:
Diagnostic Test: ultrasound — trans-vaginal and trans-abdominal ultrasound using different modalities such as grey-scale, Doppler, multi-planer mode
Procedure: closure of uterine wall defect — uterine incision above placental bulge by at least 5 mm then complete separation of the placenta starting from areas of least resistance to areas of high resistance leaving a clear defect which will be closed by non locked running sutures from inside the uterus starting from one edge, hitch the bed to the other edge of the defect and controlling placental bed hemorrhage then closing the uterine incision via running sutures in 2 layers with compressing the bed from outwards in the first layer. hemostasis of the abnormal pelvic vasculature if excessive bleeding internal iliac artery may be ligated then insertion of intra-peritoneal drain followed by closing the abdomen.
  Other Names: Double compression suture

SUMMARY:
participants diagnosed as placenta accreta spectrum were subjected to cesarean delivery.

Investigators manually detected a plan of cleavage through which the placenta was separated followed by closure of defective placental bed.

Data were collected about the outcome.

DETAILED DESCRIPTION:
Demographic data, detailed history taking, routine blood tests were done. Trans-abdominal and trans-vaginal ultrasound to diagnose placenta accreta spectrum ( PAS). Detecting new signs to help sure diagnosis of PAS.

Cesarean section will be performed through extended transverse supra-pubic incision bladder dissection from anterior uterine wall using electro-coagulation instruments and double ligation of large caliber bridging vessels.

Uterine incision above the placental bulge by at least 5 mm then complete separation of the placenta starting from least resistance plans to high resistant one leaving a clear defect which will be closed by running sutures from inside the uterus and controlling placental bed hemorrhage then closing the uterine incision with compressing the bed from outwards ( double compression sutures ) internal Iliac artery ligation may be done as a complementary measure to control the bleeding from abnormal pelvic vasculature, insertion of intraperitoneal drain and closure of abdominal wall in layers.

ELIGIBILITY:
Inclusion Criteria:

* pregnant women diagnosed as placenta accreta spectrum with previous Cesarean section, with or without other uterine surgeries and less than 40 years of age.

Exclusion Criteria:

* pregnant women having medical conditions such as cardiac diseases, coagulopathy and hematological disorders.

pregnant women had 5 or more previous Cesarean sections or their age more than 40 years

Ages: 19 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 159 (Actual)
Dates: Start 2020-07-28 (Actual); Primary Completion 2023-04-20 (Actual); Study Completion 2023-05-20 (Actual)

PRIMARY OUTCOMES:
surgical outcome | from the time of the surgery until 48 hours after.
  number of participants whom their uterus were preserved without major hemorrhage
intra-operative blood loss | intraoperative
  the amount of blood loss during operation was estimated for each participant.
surgical complications | intraoperative
  number of participants had bladder, ureter injury or hysterectomy,
internal iliac artery ligation | intra-operative
  number of participants had with either unilateral or bilateral internal iliac artery ligation
high dependency unit admission | from 0 to 48 hours postoperative
  number of participants needed high dependency unit admission
wound complications | up to 2 weeks postoperative
  number of patients suffered wound infection
change in the hemoglobin level | from 48 hours pre operative to 48 hours post operative
  participant's hemoglobin was measured
blood transfusion | from 48 hours preoperative to 48 hours postoperative.
  number of units of blood and it's products transfused to participants
hematuria | post-operative up to 24 hours
  number of participants suffered hematuria
manual cervical assesment | before skin incision
  participants were subjected to vaginal examination to asses the cervix lenght
placental separation | intra-operative
  number of participants whom their placenta was separated manually
surgical grading of the placenta | intra-operative
  number of participants who had accreta, increta, percreta or mixed type
ultrasound grading of the placenta | pre-operative
  number of participants who were diagnosed by ultrasound as accreta, increta or percreta
manual assessment of vaginal fornices | before skin incision
  participants were subjected to vaginal examination to assess fornices
repair time | intra-operative
  the time recorded from the end of the placental separation to the closure of the first layer of the uterus
total operation time | intra-operative
  the time taken from the start of the skin incision to the skin closure

SECONDARY OUTCOMES:
placental bed | intra-operative
  number of participants that investigators detected a well delineated placental bed like a pouch
pouch site | intra-operative
  the site of the pouch in relation to the cervix
defect site | intra-operative
  the location of the myometrium defects

OTHER OUTCOMES:
new ultrasound sign the pouch | pre-operative
  number of participants that the investigators detected the previously noticed pouch by ultrasound.
significance of the pouch | peri-operative
  the investigators determine the relation of the pouch to estimated blood loss
Pathology | From the operation time for 48 hours
  Histopathological examination of 1 cm specimen from the myometriam attached to the placenta in random cases

CONTACTS AND LOCATIONS:
Overall Officials: Mahmoud AH Hamdy, A. lecturer, Principal Investigator — faculty of medicine department of obstetrics and gyneacology
Locations (1):
- Faculty of Medicine, Alexandria, Egypt

IPD SHARING:
Plan to Share IPD: Yes
all IPD that underlies results in publication
Supporting Information: Study Protocol
Time Frame: after publication by 1 month

REFERENCES:
- [Result] Sentilhes L, Kayem G, Chandraharan E, Palacios-Jaraquemada J, Jauniaux E; FIGO Placenta Accreta Diagnosis and Management Expert Consensus Panel. FIGO consensus guidelines on placenta accreta spectrum disorders: Conservative management. Int J Gynaecol Obstet. 2018 Mar;140(3):291-298. doi: 10.1002/ijgo.12410. No abstract available. PMID 29405320